CLINICAL TRIAL: NCT04572984
Title: The Study for Diagnostic Value and Safety of Transbronchial Mediastinal Cryobiopsy Combined With EBUS-TBNA in Mediastinal Lesions
Brief Title: Transbronchial Mediastinal Cryobiopsy Combined With EBUS-TBNA in the Diagnosis of Mediastinal Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Third Military Medical University (Other)
Collaborators: Heidelberg University (Other)
Responsible Party: Principal Investigator, Ye Fan, Principal Investigator, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: EBUS-TBMCB 2020
Record Dates: First submitted 2020-09-12; First posted 2020-10-05 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Mediastinal Lymphadenopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EBUS-TBNA-TBMCB (Experimental): endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) was followed by endobronchial ultrasound-guided transbronchial mediastinal cryobiopsy (EBUS-TBMCB)
  Interventions: Procedure: EBUS-TBMCB
- EBUS-TBNA (No Intervention): endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) was performed

INTERVENTIONS:
Procedure: EBUS-TBMCB — endobronchial ultrasound-guided transbronchial mediastinal cryobiopsy was performed in experimental arm following EBUS-TBNA
  Arms: EBUS-TBNA-TBMCB

SUMMARY:
The clinical study is aimed to prospectively evaluate the diagnostic accuracy and the safety of adding transbronchial mediastinal cryobiopsy to standard sampling in mediastinal diseases.

DETAILED DESCRIPTION:
A traditional method, endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) was used to be compared. The patients involved were randomly divided into two groups. In the experimental group, EBUS-TBMCB was performed following EBUS-TBNA while in the other group, EBUS-TBNA was performed respectively. The samples obtained in the two groups were analyzed by the pathologists. Patients were followed up for confirming the diagnosis and complications. The diagnostic accuracy and prevalence of procedure-related adverse events were compared between the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Age >=15 years;
* More than one mediastinal lesions with diameter >= 1cm was detected by thoracic CT;
* Indication of biopsy to identify the etiology, including recently discovered mediastinal lesions or combination of clinical respiratory symptoms and complicated lung lesions implicated by thoracic image ;
* Completion of necessary preoperative laboratory examination and other examinations such as cardiac ultrasound or CTA when necessary, in order to exclude potential contradictions;
* Informed consent form achievement.

Exclusion Criteria:

* Contradictions to bronchoscopy examination such as severe cardiopulmonary diseases, coagulation disorders, intolerance to anesthesia or endoscopic operation and so on;
* Failure to detect the mediastinal lesions in ultrasonic landscape;
* Cysts or abscess;
* Requirements for additional procedures other than EBUS examination (such as endobronchial biopsy);
* Psychiatric disorders or severe neurosis.
* Participation in other clinical experiments in recent 3 months;
* Any other conditions considered to be inappropriate to be involved in this study.

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
diagnostic yield | through study completion, an average of 1 year
  percentage of patients for whom the EBUS procedures provided a definite diagnosis in each arm
prevalence of the procedure-related adverse events | through study completion, an average of 1 year
  the ratio of the number of patients who had adverse events caused by the procedure and the number of all the patients who have undergone this procedure in each arm

SECONDARY OUTCOMES:
sample size | through study completion, an average of 1 year
  the area and diameter of sample obtained by each procedure
consumed time | through study completion, an average of 1 year
  duration of each period in each procedure
sample adequacy | through study completion, an average of 1 year
  the ratio of the number of patients with adequate sample by the procedure and the number of all the patients who have undergone this procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ye Fan, PhD, Principal Investigator — Third Military Medical University; Felix Herth, Principal Investigator — Thoraxklinik - Heidelberg University Hospital
Locations (2):
- The Army Medical University, Chongqing, Chongqing Municipality, China
- Thoraxklinik - Heidelberg University Hospital, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fan Y, Zhang AM, Wu XL, Huang ZS, Kontogianni K, Sun K, Fu WL, Wu N, Kuebler WM, Herth FJF. Transbronchial needle aspiration combined with cryobiopsy in the diagnosis of mediastinal diseases: a multicentre, open-label, randomised trial. Lancet Respir Med. 2023 Mar;11(3):256-264. doi: 10.1016/S2213-2600(22)00392-7. Epub 2022 Oct 22. PMID 36279880

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT04572984/Prot_SAP_002.pdf